CLINICAL TRIAL: NCT00683306
Title: Multicentre, Open Label, Extension Study of Treatment With Gefitinib(IRESSA™) for Patients Completing Other Gefitinib Clinical Studies Who May Benefit From Gefitinib Treatment
Brief Title: Open Label Extension Study With Gefitinib (IRESSA™) for Completing Trial Patients Who May Benefit From Further Treatment
Status: Approved for marketing | Type: Expanded Access
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D791AC00008
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-08

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: ZD1839 (Iressa) — Gefitinib supplied for oral use at the dose and schedule that the patient received in the previous gefitinib clinical study. In the case of placebo patients, the gefitinib dose will be as described in the protocol of their previous gefitinib clinical study.
  Other Names: Iressa

SUMMARY:
The purpose of this study is to provide gefitinib treatment to patients who, on completion or closure of other gefitinib clinical studies, were either receiving placebo treatment, or are continuing on the same dose and regimen of gefitinib established in their preceding study, for as long as the patients continue to derive benefit.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed preceding gefitinib therapy from either the 1839IL/0709 (250mg dosing) study or 1839IL/0710 (250mg dosing) study and in the opinion of the investigator may benefit from further gefitinib treatment.
* No more than 14 days lapse in gefitinib treatment between the patient completing the preceding gefitinib clinical study and beginning of this study except when agreed by the AstraZeneca physician.

Exclusion Criteria:

* Any evidence of clinically active interstitial lung disease (patients with chronic,stable, radiographic changes who are asymptomatic need not be excluded).
* In the opinion of the investigator, any evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease).
* Withdrawal, at any time, from the preceding gefitinib study.
* Concomitant use of phenytoin, carbamazepine, rifampicin, barbiturates, or St John's Wort

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Rukazenkov, Study Director — AstraZeneca
Locations (54):
- Research Site, La Plata, Argentina
- Research Site, Concord, Australia
- Austria (3):
  - Research Site, Graz
  - Research Site, Linz
  - Research Site, Vienna
- Brazil (5):
  - Research Site, Fortaleza
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
  - Research Site, Sorocaba
- Bulgaria (4):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Deszk
  - Research Site, Mosdós
  - Research Site, Pécs
  - Research Site, Zalaegerszeg
- India (7):
  - Research Site, Hyderabad
  - Research Site, Karnataka
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Vellore
- Latvia (2):
  - Research Site, Daugavpils
  - Research Site, Riga
- Malaysia (3):
  - Research Site, George Town
  - Research Site, Kampung Baharu Nilai
  - Research Site, Kuala Lumpur
- Mexico (4):
  - Research Site, Durango
  - Research Site, Mexico City
  - Research Site, Monterrey
  - Research Site, Torreón
- Philippines (3):
  - Research Site, Manila
  - Research Site, Pasig
  - Research Site, Quezon City
- Romania (2):
  - Research Site, Bucharest
  - Research Site, Iași
- Research Site, Moscow, Russia
- Research Site, Singapore, Singapore
- Research Site, Johannesburg, South Africa
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (2):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
- Turkey (Türkiye) (2):
  - Research Site, Ankara
  - Research Site, Istanbul